CLINICAL TRIAL: NCT05651152
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Nighttime Doses of JZP441 in Sleep-Deprived Healthy Participants: A Double-Blind, Randomized, Placebo-Controlled Phase 1 Study
Brief Title: A Study to Investigate The Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JZP441 in Sleep-deprived Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JZP441-101
Record Dates: First submitted 2022-11-28; First posted 2022-12-14 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; JZP441

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind (participants and site staff [excluding site pharmacy staff])
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JZP441 (Experimental): Participants who will be randomized to receive an oral dose of JZP441.
  Interventions: Drug: JZP441
- Placebo (Placebo Comparator): Participants who will be randomized to receive an oral dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JZP441 — Nighttime oral dose
  Arms: JZP441
Drug: Placebo — Nighttime oral dose
  Arms: Placebo

SUMMARY:
This Phase 1, double-blind, randomized, placebo-controlled study will characterize the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of ascending nighttime doses of JZP441 in sleep-deprived healthy participants.

DETAILED DESCRIPTION:
This study will initially employ nighttime dosing in sleep-deprived healthy participants. Participants (up to 12 per cohort) will be randomized to study intervention. Participants will remain awake during the day and then will be dosed at night. Safety, tolerability, PK and PD assessments will be conducted for nighttime dose.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age inclusive, at the time of signing the informed consent
* Are overtly healthy as determined by medical evaluation, including medical history, physical exam, laboratory tests, and cardiac/blood pressure monitoring

Exclusion Criteria:

* Female participants who are pregnant, nursing, or lactating
* History or presence of clinically significant allergy or allergy to band aids, adhesive dressing, electrocardiogram (ECG) patches, or medical tape
* History or presence of gastrointestinal (including prior bariatric bypass surgery), hepatic or renal disease, or any other condition that may interfere with absorption, distribution, metabolism, or excretion of drugs
* Presence of renal impairment or calculated creatinine clearance < 80 mL/min
* Triplicate 12-lead ECG demonstrating a mean QTcF > 450 msec for males and > 470 msec for females or any other clinically significant ECG abnormality per investigator assessment at Screening or Day -1
* Presence or history of significant cardiovascular disease including but not limited to: myocardial infarction, uncontrolled hypertension, systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg (at Screening or Day -1), angina pectoris, clinically significant arrhythmias, clinically significant valvular heart disease, history of any revascularization procedures or second or third-degree heart block with/without a pacemaker, heart failure, or family history of Torsades de Pointes
* Laboratory value(s) outside the laboratory reference range that are considered to be clinically significant by the investigator
* Current diagnosis of or receiving treatment for depression; past (within 5 years) major depressive episode according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) criteria; history of suicide attempt, current suicidal risk as determined from history, or presence of active suicidal ideation
* History or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to DSM-5 criteria
* Participation in another clinical study of an investigational drug or medical device within 30 days or 5 half-lives (whichever is longer) prior to check-in on Day -1
* Presence at Screening of human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis C antibody, or a clinical history of these infections
* History of chronic insomnia (as defined by DSM-5 criteria)
* Has been diagnosed with sleep apnea or been identified as being at high risk for sleep apnea by standardized questionnaire (STOP-BANG)
* Any clinically relevant medical, behavioral, or psychiatric disorder that is associated with excessive sleepiness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events After Administration of JZP441 in Sleep-deprived Healthy Participants | 1 hour postdose up to Day 8

SECONDARY OUTCOMES:
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) Levels of JZP441 | Pre-dose and multiple post-dose timepoints, up to 36 hours
Pharmacokinetic Parameter Time to Maximum Plasma Concentration (Tmax) of JZP441 | Pre-dose and multiple post-dose timepoints, up to 36 hours
Pharmacokinetic Parameter Area Under the Concentration-Time Curve (AUC) of JZP441 | Pre-dose and multiple post-dose timepoints, up to 36 hours

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Site 1, Eatontown, New Jersey
  - Clinical Site 2, New York, New York